CLINICAL TRIAL: NCT02080039
Title: Clinical Pilot Study of the Effect of Electrical Stimulation of Denervated Muscles After Spinal Cord Injury
Brief Title: Electrical Stimulation of Denervated Muscles After Spinal Cord Injury
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-13
Record Dates: First submitted 2014-02-24; First posted 2014-03-06 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Spinal Cord Injury
Keywords: Spinal Cord Injury; Denervation; Electrical Stimulation
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Electric Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Electrical Stimulation (Experimental)
  Interventions: Device: Electrical Stimulation

INTERVENTIONS:
Device: Electrical Stimulation

SUMMARY:
In this study the following hypotheses will be tested:

Electrical stimulation of the gluteal muscle (buttocks) leads to

1. an increase in the thickness of the gluteal muscle
2. a decrease in the thickness of the fat of the buttock area
3. a change in the distribution of the middle and maximal seating pressure to a more consistent pressure
4. an increase in well-being of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Duration of palsy: minimum two years after traumatic or non-traumatic spinal cord injury
* Level of lesion: T 10 to L 5, AIS A, classified by the American Spinal Injury Association (AISA)

Exclusion Criteria:

* Acute decubitus in the stimulated area
* Arteriosclerosis
* Less than three months after flap surgery or after decubitus in the stimulated area
* Infections or skin eczema in the stimulated area

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-09; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Magnetic Resonance Imaging to determine the thickness of the gluteal muscle and fat tissue of the buttock. | 45 min.

SECONDARY OUTCOMES:
Measuring of the seating pressure to determine the distribution of the middle and maximal seating pressure | 15 min.
Questionnaire on subjective wellbeing | 10 min.
  The subjective effect of the electric stimulation will be assessed by an 5-item-questionnaire. Since no standardised questionnaire is available to assess the well-being in relation to sitting in a wheelchair, an individual non-validated questionnaire has been developed. It contains five questions: Question 1 and 2 address the number of resting phases while lying down and the respective overall duration of decompression each day. The questions 3 to 5 focus on the fear of pressure sores while sitting, every day limitations based on decompression phases and the subjective well-being while sitting in a wheelchair. The subjects answer the questions using a visual analog scale of 10 cm, indicating 0=no fear/no impairment/no well-being; 10=high fear/high impairment/high well-being. The subjects complete the questionnaire at baseline (start of intervention), after three and after six months.

CONTACTS AND LOCATIONS:
Locations (1):
- Swiss Paraplegic Centre, Nottwil, Canton of Lucerne, Switzerland